CLINICAL TRIAL: NCT04656015
Title: Cardiovascular Manifestation of Inflamatory Bowel Disease Patient ( Tissue Doppler Echocardiography and Cardiac MRI )
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mervat Sayed Kamal Sayed, resident doctor, Assiut University
Other Study IDs: cardiac MRI in IBD patient
Record Dates: First submitted 2020-11-23; First posted 2020-12-07 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-11

CONDITIONS: Cardiac MRI in IBD Patient

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRI — cMRI will be done only to patients presented with signs of HF, with raised cardiac biomarkers and echocardiographic signs of myocardial injury
  The Lake Louise diagnostic criteria for CMR in myocarditis:
  CMR findings are consistent with myocardial inflammation if at least two of the following criteria are present:
  * Regional or global myocardial signal intensity increase in T2-weighted images
  * Increased global myocardial early gadolinium enhancement ratio between myocardium and skeletal muscle in gadolinium-enhanced T1-weighted images
  * There is at least one focal lesion with non-ischemic regional distribution on late gadolinium enhancement Presence of left ventricular dysfunction or pericardial effusion provides additional, supportive evidence for myocarditis 6. Carotid du

SUMMARY:
1. Evaluation of cardiovascular changes using Doppler echocardiography and cardiac MRI in IBD patients
2. To detect the frequency of myocardial injury in IBD patients
3. To detect the sensitivity and specificity of echocardiography for the detection of cardiac injury in comparison to cardiac MRI in IBD patients

DETAILED DESCRIPTION:
The burden of extra-intestinal disease is high in patients with IBD, some of whom respond to or are prevented by treating the bowel inflammation, whereas others require specific treatment because they are independent of the underlying bowel inflammation .

Cardiovascular diseases are the major causes of mortality and morbidity worldwide. They may arise for various reasons such as obesity, type 2 diabetes, genetic, environmental, dietary, and lifestyle factors. Besides all these, there is much evidence suggesting that inflammation is an important player in the pathogenesis of heart disease, as well as atherogenesis and atherosclerosis . A most common systemic inflammatory disease is inflammatory bowel disease (IBD), which is a collection of ulcerative colitis and Crohn's disease, a chronic intestinal disease that may arise due to different factors, and is precipitated by environmental and genetic susceptibility Tissue Doppler imaging (TDI) is a useful echocardiographic technique to evaluate global and regional myocardial systolic as well as diastolic function. It can also be used to quantify right ventricular and left atrial function.

To date, cardiac magnetic resonance imaging (cMRI) is mostly used to detect significantly decreased EFs and abnormalities in wall motion. Contrast enhancement (CE) CMR is a more sensitive technique of cMRI and can detect areas of myocardial damage in patients with acute myocarditis .

ELIGIBILITY:
Inclusion Criteria:

* IBD patients presented with disease flare, which is grouped by the 3 domains of disease severity:

  * Measurable inflammatory burden (C-reactive protein, mucosal lesions, upper gastrointestinal involvement, and disease extent.
  * Disease course (including structural damage, history/extension of intestinal resection, perianal disease, number of flares, and extraintestinal manifestations)

Exclusion Criteria:

* Patients with poor echocardiographic window, previously diagnosed as IHD, complete heart block, mitral stenosis, prosthetic mitral valve, congenital heart disease with a left to right shunt, and CKD patients will be excluded from the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: IBD patients presented with disease flare, which is grouped by the 3 domains of disease severity:
  * Measurable inflammatory burden (C-reactive protein, mucosal lesions, upper gastrointestinal involvement, and disease extent.
  * Disease course (including structural damage, history/extension of intestinal resection, perianal disease, number of flares, and extraintestinal manifestations)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of cardiovascular affection in IBD patients | baseline
  Incidence of cardiovascular affection in IBD patients

SECONDARY OUTCOMES:
Incidence of cardiovascular affection in IBD patients | baseline
  Incidence of cardiovascular affection in IBD patients

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Mohamed, Principal Investigator — Assiut univerty

REFERENCES:
- [Background] Bernstein CN, Benchimol EI, Bitton A, Murthy SK, Nguyen GC, Lee K, Cooke-Lauder J, Kaplan GG. The Impact of Inflammatory Bowel Disease in Canada 2018: Extra-intestinal Diseases in IBD. J Can Assoc Gastroenterol. 2019 Feb;2(Suppl 1):S73-S80. doi: 10.1093/jcag/gwy053. Epub 2018 Nov 2. PMID 31294387
- [Background] Matsuura E, Atzeni F, Sarzi-Puttini P, Turiel M, Lopez LR, Nurmohamed MT. Is atherosclerosis an autoimmune disease? BMC Med. 2014 Mar 18;12:47. doi: 10.1186/1741-7015-12-47. PMID 24642015
- [Background] Fung G, Luo H, Qiu Y, Yang D, McManus B. Myocarditis. Circ Res. 2016 Feb 5;118(3):496-514. doi: 10.1161/CIRCRESAHA.115.306573. PMID 26846643